CLINICAL TRIAL: NCT06978361
Title: Comparison of Efficacy of Microneedling With Autologous Platelet-Rich Plasma vs Microneedling With Topical Insulin in the Treatment of Atrophic Acne Scars
Brief Title: Comparison of Efficacy of Microneedling With Platelet Rich Plasma Vs Microneedling With Topical Insulin in the Treatment of Acne Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Khyber Teaching Hospital (Other)
Responsible Party: Principal Investigator, Soaiba Naeem, Doctor, Khyber Teaching Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 938/DME/KMC
Record Dates: First submitted 2025-05-10; First posted 2025-05-18 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-02

CONDITIONS: Post-acne Atrophic Scars
Keywords: Post-acne atrophic scars; Microneedling with autologous Platelet- Rich Plasma; Microneedling with topical insulin
MeSH Terms: interventions — Percutaneous Collagen Induction; Insulin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A , Microneedling with autologous PRP (Experimental): Patients in group A will undergo microneedling with autologous PRP i.e cleansing of the treatment area with an antiseptic solution will be performed.Topical anesthetic will be applied to the area for 20-30 mins .Approximately 10ml of blood will be drawn into sterile tubes. blood sample will be placed in centrifuge 10-15mins which separates the blood components, allowing for the collection of PRP .Then sterile microneedling device will be used to begin the procedure by adjusting the needle depth according to scar severity.Controlled microinjuries to the skin will be made by moving the device in a systematic pattern over the treatment area .After microneedling ,immediately harvested PRP will be applied to the treated area ,allowing it to penetrate into the microinjuries .Patient will be asked for consideration of aftercare instructions ,including avoiding sun exposure , harsh skincare products and strenuous exercise for few days.
  Interventions: Procedure: Microneedling with autologous Platelet Rich Plasma
- Group B , Microneedling with Topical insulin (Experimental): Patients in group B will undergo microneedling with Topical insulin i.e cleansing of the treatment area with an antiseptic solution will be performed.Topical anesthetic will be applied to the area for 20-30 mins to reduce discomfort during the procedure.Then sterile microneedling device will be used to begin the procedure by adjusting the needle depth according to scar severity.Controlled microinjuries to the skin will be made by moving the device in a systematic pattern over the treatment area .After microneedling Insulin (Regular) will be applied immediately to the treated area. insulin will be allowed to penetrate into the microinjuries created by the microneedling for about 30 mins . Patient will be asked for consideration of aftercare instructions ,including avoiding sun exposure , harsh skincare products and strenuous exercise for few days.
  Interventions: Procedure: Microneedling with topical insulin

INTERVENTIONS:
Procedure: Microneedling with autologous Platelet Rich Plasma — Patients in group A will undergo Microneedling with autologous PRP
  Arms: Group A , Microneedling with autologous PRP
Procedure: Microneedling with topical insulin — Patients in group B will undergo Microneedling with Topical insulin ( regular).
  Arms: Group B , Microneedling with Topical insulin

SUMMARY:
This study compares the outcome of two procedures for the treatment of atrophic acne scars.

DETAILED DESCRIPTION:
Post acne scars develop due to severely inflamed and nodulocystic acne. Numerous methods exist for the treatment of post acne scars including lasers , microneedling and chemical peels etc . This study is to compare the efficacy two procedures.

ELIGIBILITY:
Inclusion Criteria:

Patients confirmed with post-acne atrophic scars . No prior treatment for scars in last 6 months.

-

Exclusion Criteria:

* Patient with active acne or other skin conditions (e.g eczema , psoriasis). Patients on oral or topical retinoids. Pregnant or lactating Mothers. Patients with recurrent herpes simplex infection. Previous Hx of keloids / hypertrophic scarring. Deranged blood glucose levels. Bleeding disorders

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy of treatment | 6 months
  Efficacy will be determined by using the Goodman and Baron's Scarring Grading System as" Percentage of decrease in acne scar grade" i.e calculated through subtracting post treatment grade from pre treatment grade and then multiplying it with 100 in both treatment groups .

CONTACTS AND LOCATIONS:
Locations (1):
- Khyber Teaching Hospital, Peshawar, KPK ,Pakistan, Pakistan

IPD SHARING:
Plan to Share IPD: No
Patient's confidentiality may be breached .